CLINICAL TRIAL: NCT06980792
Title: Surgical Approach for Adenocarcinoma of the Pancreas With Synchronous Liver Metastases
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Fabrizio Di Benedetto, Professor of Surgery, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 396/2021/OSS/AOUMO; ISLS pancreas study group (Other: ISLS)
Record Dates: First submitted 2025-04-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Neoplasms; Liver Metastasis; Pancreas Ductal Adenocarcinoma; Surgery of the Pancreatic Head; Liver Resection; Pancreatectomy
Keywords: PDAC; MIPS; whipple; distal pancreatectomy; RAMPS; hepatectomy; liver resection; metastasis; metastases; synchronous; ISLS
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Pancreatectomy; Hepatectomy; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical group: Patients that underwent pancreatic and liver surgery
  Interventions: Procedure: Pancreatectomy and liver resection
- Non-surgical group: Patients that underwent CHT alone
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Pancreatectomy and liver resection — Surgery for synchronous liver metastasis from PDAC with or without previous neoadjuvant chemotherapy
  Groups: Surgical group
Drug: Chemotherapy — Chemotherapy alone in potentially resectable patients with PDAC and synchronous liver metastasis
  Groups: Non-surgical group

SUMMARY:
The study focuses on patients with synchronous liver metastasis from pancreatic adenocarcinoma that underwent both pancreatic and liver resection. The control group is made up of patients with resectable or borderline resectable pancreatic adenocarcinoma and synchronous liver metastasis that were excluded from surgery. Short and long-term outcomes will be compared to evaluate the safety and efficacy of simultaneous liver and pancreatic resection.

DETAILED DESCRIPTION:
1. Summary:

   The study focuses on patients with synchronous liver metastasis from pancreatic adenocarcinoma that underwent both pancreatic and liver resection. The control group is made up of patients with resectable or borderline resectable pancreatic adenocarcinoma and synchronous liver metastasis that were excluded from surgery. Short and long-term outcomes will be compared to evaluate the safety and efficacy of simultaneous liver and pancreatic resection.
2. Introduction 2.1 Background and rationale The most common pathological pattern of pancreatic tumor is pancreatic ductal adenocarcinoma (PDAC), which accounts for approximately 90% of all cases. For digestive tract tumors such as colorectal, gastric, and pancreatic tumors, distant metastases often represent the last stage of the disease evolvement, and liver is a frequent disseminate site for metastatic tumor. Among them, only hepatic resection for metastatic disease has gained general acceptance as a potentially curative option in patients with colorectal cancer. The role of surgery for metastases from neuroendocrine tumors on long-term outcome is also well-documented. Recently, Markar et al. reported that surgical resection of hepatic metastases from gastric adenocarcinoma was associated with a significantly improved overall survival (p < 0.001). Moreover, they confirmed the additional survival benefit of solitary compared with multiple hepatic metastases (odds ratio = 0.31; p = 0.011). Liver resection showed longer survival rates also for pancreatic neuroendocrine tumor (PNET) patients.

   However, historical results regarding hepatic resection for PDAC were in conflicts and remained controversial. Furthermore, rare systematic review or meta-analysis was ever reported focusing on PDAC as a separate group. A recent meta-analysis reported that overall survival of PDAC patients can benefit from hepatic resection to some extent. It has been also recently showed that that surgical resection of pancreatic cancer with synchronous liver oligometastases is safe, and it can be associated with improved survival, providing a careful selection of patients after primary chemotherapy. Since a randomized controlled trial may be ethically questionable, a multicenter international retrospective study may clarify the role of liver resection in this cohort of patients.

   2.2 Objectives

   The primary aim is to examine recurrence free survival (RFS) and overall survival (OS) following surgical resection of synchronous hepatic metastases from PDAC, and to study the role of tumor burden and chemotherapy regimen on survival.
3. Methods:

3.1 Study design Patients underwent liver resection for synchronous metastases from pancreatic adenocarcinoma, single or multiple metastasis, will be included in the study, without any time interval limitation.

Clinical features, operative data and chemotherapy regimens will be analyzed. A control group of non-surgical patients will be included in the study for a propensity score match.

3.2 Setting

* No time interval limitation for recruitment
* No volume-based restriction for center eligibility 3.3 Participants Patients of age >18, underwent surgery for pancreatic adenocarcinoma (duodenopancreatectomy, distal pancreatectomy, total pancreatectomy) and liver resection (major or minor) for synchronous metastasis, that received neoadjuvant and/or adjuvant chemotherapy. The control group is made up of patients age >18 with resectable or borderline resectable pancreatic adenocarcinoma and synchronous liver metastasis that didn't underwent surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age >18, underwent surgery for pancreatic adenocarcinoma (duodenopancreatectomy, distal pancreatectomy, total pancreatectomy) and liver resection (major or minor) for synchronous metastasis, that received neoadjuvant and/or adjuvant chemotherapy.
* The control group is made up of patients age >18 with resectable or borderline resectable pancreatic adenocarcinoma and synchronous liver metastasis that didn't underwent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent liver resection for synchronous metastases from pancreatic adenocarcinoma, single or multiple metastasis, will be included in the study, without any time interval limitation. Clinical features, operative data and chemotherapy regimens will be analyzed. A control group of non-surgical patients will be included in the study for a propensity score match. Setting
  * No time interval limitation for recruitment
  * No volume-based restriction for center eligibility
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
Recurrence-free survival | 3 years

SECONDARY OUTCOMES:
Post-operative short-term outcomes 1 | 90 days
  comprehensive complication index (using the online official CCI calculator that combines the events based on the Clavien-Dindo Classification)

OTHER OUTCOMES:
Post-operative short-term outcomes 2 | up to 100 weeks
  ICU and in-hospital stay (days)
Post-operative short-term outcomes 3 (histology) | up to 100 weeks
  surgical margin (in millimeters) and R status (R 0: no infiltration; R 1: microscopic infiltration; R 2: macroscopic infiltration) of pancreatic and hepatic specimens; nodal status (number of nodes sampled and number of positive nodes)

CONTACTS AND LOCATIONS:
Locations (1):
- AOU di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided